CLINICAL TRIAL: NCT02932293
Title: Triple Combination DAAs for Ultra Short Duration Therapy for HCV Genotype 1b in Chinese (SODAPI II Study)
Brief Title: Triple Combination DAAs for Treating HCV GT1b Subjects
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The collaborating pharmaceutical company will not wish to continue with the trial due to the internal issues in the company.
Sponsor: Humanity and Health Research Centre (Other)
Collaborators: University of Maryland (Other); Emory University (Other); Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H&H_SODAPI II
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2016-10

CONDITIONS: Chronic Hepatitis C Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF+DCV+SMV 3-4 wks (Experimental): Patients without cirrhosis will receive sofosbuvir, daclatasvir and simeprevir for (a) 3 weeks if HCV viral load on day 2 is <500 IU/ml or (b) 4 weeks if HCV viral load on day 2 is >500 IU/ml.
  Interventions: Drug: SOF+DCV+SMV
- SOF+DCV+SMV 6-8 wks (Experimental): Patients with cirrhosis and CP-A will receive sofosbuvir, daclatasvir and simeprevir (a) 6 weeks if HCV VL on day 2 is <500 IU/ml or (b) 8 weeks if HCV VL on day 2 is >500 IU/ml.
  Interventions: Drug: SOF+DCV+SMV

INTERVENTIONS:
Drug: SOF+DCV+SMV — Sofosbuvir (SOF) 400 mg tablet administered orally once daily; Daclatasvir (DCV) 60 mg tablet administered orally once daily; Simeprevir (SMV) 150 mg tablet orally once daily.

SUMMARY:
There is only one kind of treatment (simeprevir 150 mg + sofosbuvir 400 mg+daclatasvir 60 mg) in this study but the treatment duration may be different depending on patients' response to the antiviral therapy and whether patients have liver cirrhosis. If patients have no cirrhosis and the HCV viral load on day 2 is <500 IU/ml, patients will receive sofosbuvir, daclatasvir and simeprevir for 3 weeks, otherwise the treatment duration is 4 weeks. If patients have cirrhosis and the HCV viral load on day 2 is <500 IU/ml, patients will receive sofosbuvir, daclatasvir and simeprevir for 6 weeks, otherwise the treatment duration will be 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. HCV RNA positive >2000 IU/ml or NAT POC positive
2. Genotype 1b
3. CP score ≤6

Exclusion Criteria:

1. Pregnant or nursing female or male with pregnant female partner
2. Hematologic or biochemical parameters at Screening outside the protocol- specified requirements
3. Active or recent history (≤ 1 year) of drug or alcohol abuse
4. Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers)
5. History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with plasma HCV viral load below the lower limit of quantification for 12 weeks after treatment completion (SVR12) | Post treatment Week 12
  SVR12 is defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after last dose of study drug.

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Baseline up to Week 24
Proportion of participants with unquantifiable HCV viral load at specified time points during and after treatment | Baseline up to Week 24
Kinetics of circulating HCV RNA during treatment and after treatment discontinuation | Baseline up to Week 24
Proportion of participants with on-treatment virologic breakthrough and relapse | Baseline up to Week 24
  Viral breakthrough is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) during treatment, but did not achieve a sustained virologic response (SVR). Viral relapse is defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) within 4 weeks of end of treatment, but did not achieve an SVR up to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: George LAU, MD, Principal Investigator — Humanity & Health Medical Centre
Locations (1):
- Humanity and Health Medical Centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided